CLINICAL TRIAL: NCT03864133
Title: The Effects of Intraocular Phenylephrine/Ketorolac Infusion on Retinal Thickness and Macular Edema in Cataract Surgery
Brief Title: No Drop Post-Op Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00050415
Record Dates: First submitted 2019-02-13; First posted 2019-03-06 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2021-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Omidria (Other): Phenylephrine/Ketorolac (1%/0.3%) will be administered to all participants enrolled into the study.
  Interventions: Drug: Omidria

INTERVENTIONS:
Drug: Omidria — Phenylephrine and Ketorolac infusion of 1%/0.3% during cataract surgery.

SUMMARY:
This study evaluates the effect of Intraocular Phenylephrine/Ketorolac Infusion on Retinal Thickness and Macular Edema in Cataract Surgery. Participants will receive infusions of Phenylephrine/Ketorolac during surgery instead of receiving topical NSAID drops pre and post operatively.

DETAILED DESCRIPTION:
Topical NSAIDs have been known to reduce post-operative macular edema, inflammation and pain in patients undergoing cataract surgery. Routine cataract surgery without the protection of topical NSAIDs results in an increase of the number of patients with macular edema and macular thickening.

Omidria (phenylephrine and ketorolac injection 1%/0.3%) infusion is used in patients during cataract surgery to decrease post-operative pain and inflammation. It is also indicated to maintain pupil dilation during cataract surgery.

This study will evaluate whether treating patients with Omidria during cataract surgery will control post-operative pain and inflammation as well as reduce or eliminate macular edema without the use of adjunctive topical NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 55-90 years with visual significant cataracts in one or both eyes.
* Healthy individuals able to tolerate outpatient cataract surgery under local anesthesia via either phacoemulsification and/or femtosecond assisted cataract surgery. Well-controlled diabetes, hypertension will be included.
* Females of childbearing potential must agree to use a reliable method of birth control while participating in this study. Reliable methods of birth control are: abstinence, oral contraceptives, intrauterine device (IUD), DepoProvera, tubal ligation or vasectomy of the partner (with confirmed negative sperm counts) in monogamous relationship (same partner). An acceptable, although less reliable, method involves the careful use of condoms and spermicidal foam or gel and/or cervical cap or sponge. A pregnancy test is required at least 10 days from the last normal menstrual period, if the patient is a sexually active female of childbearing potential.

Exclusion Criteria:

* Allergy to Phenylephrine or NSAIDs.
* Inability to sit steady and upright for the Optical Coherence Tomography (OCT).
* Complications during surgery, including posterior capsular rupture, vitreous loss, zonular dialysis, or iris trauma.
* Macular thickness above 300 microns at baseline
* Currently taking a prostaglandin analogue
* Presence of an epiretinal membrane on the preoperative OCT.
* Retained lens fragment post-operatively.
* Inability to return for follow appointments
* Female patients who are pregnant, lactating or planning to become pregnant during the course of treatment.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Walter, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang J, Cai L, Sun Z, Ye H, Fan Q, Zhang K, Lu W, Lu Y. Risk factors for and diagnosis of pseudophakic cystoid macular edema after cataract surgery in diabetic patients. J Cataract Refract Surg. 2017 Feb;43(2):207-214. doi: 10.1016/j.jcrs.2016.11.047. PMID 28366368
- [Background] Wielders LH, Lambermont VA, Schouten JS, van den Biggelaar FJ, Worthy G, Simons RW, Winkens B, Nuijts RM. Prevention of Cystoid Macular Edema After Cataract Surgery in Nondiabetic and Diabetic Patients: A Systematic Review and Meta-Analysis. Am J Ophthalmol. 2015 Nov;160(5):968-981.e33. doi: 10.1016/j.ajo.2015.07.032. Epub 2015 Jul 29. PMID 26232601
- [Background] Novack GD. Quality of generic ophthalmic drugs. Ocul Surf. 2013 Jan;11(1):54-6. doi: 10.1016/j.jtos.2012.10.002. Epub 2012 Oct 17. No abstract available. PMID 23321360
- [Background] Kessel L, Tendal B, Jorgensen KJ, Erngaard D, Flesner P, Andresen JL, Hjortdal J. Post-cataract prevention of inflammation and macular edema by steroid and nonsteroidal anti-inflammatory eye drops: a systematic review. Ophthalmology. 2014 Oct;121(10):1915-24. doi: 10.1016/j.ophtha.2014.04.035. Epub 2014 Jun 14. PMID 24935281
- [Background] Henderson BA, Kim JY, Ament CS, Ferrufino-Ponce ZK, Grabowska A, Cremers SL. Clinical pseudophakic cystoid macular edema. Risk factors for development and duration after treatment. J Cataract Refract Surg. 2007 Sep;33(9):1550-8. doi: 10.1016/j.jcrs.2007.05.013. PMID 17720069
- [Background] Bucci FA Jr, Waterbury LD. Comparison of ketorolac 0.4% and bromfenac 0.09% at trough dosing: aqueous drug absorption and prostaglandin E2 levels. J Cataract Refract Surg. 2008 Sep;34(9):1509-12. doi: 10.1016/j.jcrs.2008.05.023. PMID 18721711
- [Background] Waterbury LD. Alternative Drug Delivery for Patients Undergoing Cataract Surgery as Demonstrated in a Canine Model. J Ocul Pharmacol Ther. 2018 Jan/Feb;34(1-2):154-160. doi: 10.1089/jop.2017.0048. Epub 2017 Dec 11. PMID 29227185
- [Background] Kim SJ, Flach AJ, Jampol LM. Nonsteroidal anti-inflammatory drugs in ophthalmology. Surv Ophthalmol. 2010 Mar-Apr;55(2):108-33. doi: 10.1016/j.survophthal.2009.07.005. PMID 20159228
- [Background] Wielders LHP, Schouten JSAG, Winkens B, van den Biggelaar FJHM, Veldhuizen CA, Findl O, Murta JCN, Goslings WRO, Tassignon MJ, Joosse MV, Henry YP, Rulo AHF, Guell JL, Amon M, Kohnen T, Nuijts RMMA; ESCRS PREMED Study Group. European multicenter trial of the prevention of cystoid macular edema after cataract surgery in nondiabetics: ESCRS PREMED study report 1. J Cataract Refract Surg. 2018 Apr;44(4):429-439. doi: 10.1016/j.jcrs.2018.01.029. PMID 29778106

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omidria
Started | 94
Completed | 94
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Omidria
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 64
  More than one race | 0
  Unknown or Not Reported | 12

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity (BCVA) (Pre-op)
Description: Best vision will be tested with lens correction using Snellen Charts.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Omidria
Number analyzed (Participants) | 94
LogMar | .28 (.2)

2. Primary Outcome: Best Corrected Visual Acuity (BCVA) (Week 2)
Description: Best vision will be tested with lens correction using Snellen Charts to determine if improvements have been made post-operatively.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Omidria
Number analyzed (Participants) | 94
LogMar | .18 (.2)

3. Primary Outcome: Best Corrected Visual Acuity (BCVA) (Week 6)
Description: Best distance vision will be measured clinically to determine if improvements have been made post-operatively.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Omidria
Number analyzed (Participants) | 94
LogMar | .11 (.2)

4. Primary Outcome: Number of Participants That Develop Presence of Cystoid Macular Edema (CME)
Description: The number of participants that develop CME will be recorded to evaluate if Omidria is sufficient in controlling CME. The presence of CME will be determined clinically.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Omidria
Number analyzed (Participants) | 94
Participants | 0

5. Primary Outcome: Change From Baseline in Macular Thickness Measurement - Number in Microns
Description: The thickness of the macula will be measured pre and post operatively using ocular imaging to determine if Omidria is sufficient in controlling thickening post-operatively - measured in number of Microns
Time Frame: Baseline and week 6
Measure: Mean (Standard Deviation); unit: Number of Microns
Arm/Group | Omidria
Number analyzed (Participants) | 94
Number of Microns | 12 (0.2)

6. Primary Outcome: Number of Participants Needing NSAID Post-operatively
Description: Need for topical NSAID (rescue med) will be assessed at all post-op visits. If at any time the patient shows signs of cystoid macular edema, inflammation or pain, NSAIDs will be administered. The number of patients needing NSAID post-operatively will help determine if NSAIDS are needed.
Time Frame: Post-op weeks 1 through 6
Measure: Count of Participants; unit: Participants
Arm/Group | Omidria
Number analyzed (Participants) | 94
Participants
  Week 1 | 0
  Week 2 | 0
  Week 3 | 0
  Week 4 | 3
  Week 5 | 0
  Week 6 | 5

7. Primary Outcome: Change in Anterior Chamber Cells From Baseline Measurement
Description: Anterior chamber cells will be assessed through a dilated eye exam to determine if NSAIDS are needed post-operatively in addition to Omidria during surgery.
  Range and meaning (if score/scale): 0-2 0 = no cell
  1. = 10-20 cells
  2. = greater than 20 cells
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: Cell Score - Score on a Scale
Arm/Group | Omidria
Number analyzed (Participants) | 94
Cell Score - Score on a Scale | .08 (0.2)

ADVERSE EVENTS:
Time Frame: Week 6
Arm/Group | Omidria
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 1/94
Other Adverse Events (participants affected / at risk) | 94/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omidria (N=94)
Blindness (Eye disorders) | 1 (1) — Blindness
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omidria (N=94)
photophobia (Eye disorders) | 94 (94) — abnormal sensitivity to light, especially of the eyes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT03864133/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT03864133/ICF_000.pdf